CLINICAL TRIAL: NCT05334537
Title: Aromaterapinin Spinal Anestezi Uygulanan Sezaryen Vakalarında Perioperatif Anksiyete Düzeyine Etkisi / The Effect Of Aromatherapy On The Level Of Intraoperative Anxiety In Caesarean Case Under Spinal Anesthesia
Brief Title: Effect of Aromatherapy on Perioperative Anxiety Level in Cesarean Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Feyza Calisir, Assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/05-14
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Midazolam Overdose; Breast Feeding
Keywords: aromatherapy; lavandula; sedative; spinal anesthesia; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Breast Feeding | interventions — Aromatherapy; almond oil

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the aromatherapy group (Experimental): After the birth of the baby, two drops of 100% pure medical lavender oil (Lavandula angustifolia) was inhaled for 5 min through an oxygen mask by groups A and C, respectively. After 5 min, 2 mg intravenous midazolam for sedation was administred to the patients who gained 1 point from the Ramsey Sedation Scale (RSS). Complications, such as nausea, vomiting, hypotension (mean arterial pressure<60 mmHg), and allergies that developed after aromatherapy, were recorded. At the end of the operation, the dose added to the initial midazolam dose for all patients and the total surgical time were recorded. VAS pain and STAI-I scores were re-evaluated at the third postoperative hour, and the satisfaction levels of each patient after aromatherapy were recorded according to the Likert scale as "very satisfied, satisfied, moderate, and not at all satisfied".
  Interventions: Other: Aromatherapy
- the control group (Placebo Comparator): Then, after the birth of the baby two drops of odorless baby oil (jojoba and almond oil) was inhaled for 5 min through an oxygen mask by groups A and C, respectively. After 5 min, 2 mg intravenous midazolam for sedation was administred to the patients who gained 1 point from the Ramsey Sedation Scale (RSS). Complications, such as nausea, vomiting, hypotension (mean arterial pressure<60 mmHg), and allergies that developed after aromatherapy, were recorded. At the end of the operation, the dose added to the initial midazolam dose for all patients and the total surgical time were recorded. VAS pain and STAI-I scores were re-evaluated at the third postoperative hour, and the satisfaction levels of each patient after aromatherapy were recorded according to the Likert scale as "very satisfied, satisfied, moderate, and not at all satisfied".
  Interventions: Other: Placebo oil (odorless baby oil- jojoba and almond oil)

INTERVENTIONS:
Other: Aromatherapy — Ninety-six patients aged between 18 and 45 years, with a height of ≥156 centimeters (cm), and a gestational age of >37 weeks, in the ASA II risk group, who were scheduled for elective CS under spinal anesthesia, were included in the study. Patients who were to undergo lavender aromatherapy with an oxygen mask after the birth of the baby were randomly divided into two groups: aromatherapy (A) (n=48) and control (C) (n=48), who inhaled odorless essential oil. Participants were admitted to the preoperative preparation room 20 min before the operation, and their age, height, weight, and ASA risk scores were recorded after their informed consent was obtained. They were monitored and sent to the operating room after their baseline anxiety levels were measured and recorded using the Visual Analog Scale (VAS) for pain and State-Trait Anxiety Inventory (STAI-I).
  Arms: the aromatherapy group
Other: Placebo oil (odorless baby oil- jojoba and almond oil) — Ninety-six patients aged between 18 and 45 years, with a height of ≥156 centimeters (cm), and a gestational age of >37 weeks, in the ASA II risk group, who were scheduled for elective CS under spinal anesthesia, were included in the study. Patients who were to undergo lavender aromatherapy with an oxygen mask after the birth of the baby were randomly divided into two groups: aromatherapy (A) (n=48) and control (C) (n=48), who inhaled odorless essential oil. Participants were admitted to the preoperative preparation room 20 min before the operation, and their age, height, weight, and ASA risk scores were recorded after their informed consent was obtained. They were monitored and sent to the operating room after their baseline anxiety levels were measured and recorded using the Visual Analog Scale (VAS) for pain and State-Trait Anxiety Inventory (STAI-I).
  Arms: the control group

SUMMARY:
Spinal anesthesia has been accepted as the first choice for elective cesarean section due to its easy application technique and elimination of the risks of difficult intubation and aspiration. Neuraxial anesthesia is considered superior to general anesthesia in terms of fetal well-being. The state of having an operation and not being aware of the operation by the patient can cause serious anxiety and fear in the patient. Fear of surgical failure, not fully understanding the anesthesia method, possible risks of anesthesia and expected pain during the postoperative recovery period contribute to the patient's anxiety. Considering the patients undergoing elective surgery under spinal anesthesia, there is a moderate level of anxiety associated with advanced age and female gender. Reducing the stress and anxiety in the patient during elective surgery will reduce the neurohormonal response to surgery and reduce complications. Early skin-to-skin contact with the mother provides many benefits to the newborn, but maternal sedation in the operating room during cesarean delivery should also be within safe limits to avoid early skin-to-skin contact. Aromatherapy relies on the use of essential oils to contribute to physical and psychological well-being. The oils can be massaged into the skin, or inhaled using a steam infusion or burner. Birth pain is a severe pain, and the feeling of pain may increase with tension, fear and anxiety during delivery. Apart from medical methods, many complementary treatments such as acupuncture, reflexology, homeopathy, hypnotherapy, music and aromatherapy are tried to reduce pain and anxiety. Lavender aromatherapy has been shown to significantly reduce anxiety or pain in various surgical procedures. There is a growing literature on the use of lavender aromatherapy as an anxiolytic agent. Based on these findings, the study aimed to contribute to early mother-to-baby contact and breast milk intake by reducing perioperative maternal anxiety and therefore the use of sedative drugs during cesarean section performed under spinal anesthesia with the intraoperative use of lavender aromatherapy. This is the first study to evaluate the effect of aromatherapy on anxiety in cases of cesarean section under anesthesia.

DETAILED DESCRIPTION:
Patients who were to undergo lavender aromatherapy with an oxygen mask after the birth of the baby were randomly divided into two groups: aromatherapy (A) (n=48) and control (C) (n=48), who inhaled odorless essential oil. Participants were admitted to the preoperative preparation room 20 min before the operation, and their age, height, weight, and ASA risk scores were recorded after their informed consent was obtained. They were monitored and sent to the operating room after their baseline anxiety levels were measured and recorded using the Visual Analog Scale (VAS) for pain and State-Trait Anxiety Inventory (STAI-I). Following local sterilization with the patient in the sitting position, the lumbar (L) region was punctured at the L3-L4 level or the L4-L5 level with a 25-G, 90 mm pencil-point spinal atraumatic needle. After visualization of the cerebral spinal fluid flow, 10 mg of 0.5% bupivacaine (Marcaine® Spinal Heavy 0.5% ampule, AstraZeneca, UK) was administered for spinal anesthesia. Then, after the birth of the baby, two drops of 100% pure medical lavender oil (Lavandula angustifolia) and two drops of odorless baby oil (jojoba and almond oil) was inhaled for 5 min through an oxygen mask by groups A and C, respectively. After 5 min, 2 mg intravenous midazolam for sedation was administred to the patients who gained 1 point from the Ramsey Sedation Scale (RSS). Complications, such as nausea, vomiting, hypotension (mean arterial pressure<60 mmHg), and allergies that developed after aromatherapy, were recorded. At the end of the operation, the dose added to the initial midazolam dose for all patients and the total surgical time were recorded. VAS pain and STAI-I scores were re-evaluated at the third postoperative hour, and the satisfaction levels of each patient after aromatherapy were recorded according to the Likert scale as "very satisfied, satisfied, moderate, and not at all satisfied".

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who underwent CS with spinal anesthesia
* Ninety-six patients aged between 18 and 45 years,
* With a height of ≥156 centimeters (cm)
* Gestational age of >37 weeks
* The American Society of Anesthesiologists (ASA) II risk group, who were scheduled for elective CS under spinal anesthesia

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Comparison between patients using aromatherapy and those without aromatherapy | Within one hour following the cesarean section
  A comparison will be made between the two groups, one group using lavender aromatherapy and one group without aromatherapy. T-tests used to assess whether the two groups are statistically different from each other. Comparisons made by comparing with the midazolam consumption. After 5 minutes from baby's birth, 2 mg intravenous midazolam for sedation was administred to the patients who gained 1 point from the Ramsey Sedation Scale. It is a six category scale that allows the evaluation of the sedation level and was created by Ramsey et al. (score 1: anxious, agitated and restless; score 2: cooperative, oriented and tranquil; score 3: responsive to commands only; score 4: brisk response to a light glabellar tap; score 5: sluggish response to a light glabellar tap or loud auditory stimulus; score 6: means no response).
Comparison between patients using aromatherapy and those without aromatherapy | Postoperative 3rd hour
  Comparison between two groups for the postoperative 3rd hour STAI-I scores. Ensuring the baby's clean breast milk intake and early mother-infant skin contact

CONTACTS AND LOCATIONS:
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No